CLINICAL TRIAL: NCT02884973
Title: Prospective Evaluation of Changes in Tissue Oxygen Saturation in Brain and Kidney in Children Admitted to Intensive Care in the Postoperative Period of Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6156
Record Dates: First submitted 2016-06-16; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-06

CONDITIONS: Congenital Heart Defect
Keywords: congenital heart; NIRS
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is estimated that the incidence of congenital heart disease varies between 0.5 and 1% of live births, 5,000 new cases per year currently in France These are serious diseases that can be life-threatening to more or less short term.

The advances in surgical techniques in recent years has improved the prognosis of these patients in the first months of life.

The success of surgery is, among other things, conditioned by a support per complex operation, involving a multimodal intensive monitoring, and respiratory and hemodynamic support techniques.

These elements of surveillance, NIRS (Near-infrared spectroscopy) allows measurement of non-invasive tissue saturation (rSO2) in cerebral and renal oxygen.

The fundamental principle of NIRS based on an estimate of the percentage proportion of cerebral oxy-hemoglobin.

A light source is emitted by NIRS and through body tissues to the brain where the light will be absorbed and refracted depending on the tissue composition in oxy-hemoglobin.

Refracted light will be analyzed by NIRS which in turn using software will help to determine a percentage of oxyhemoglobin.

Normal values of cerebral NIRS are between 50 and 80%.NIRS can be used according to this principle to estimate cerebral tissue oxygenation but also for other tissues such as the kidney.

More than the figure, those are changes NIRS compared to a baseline that will alert us to the conditions of tissue oxygenation and allow us to identify hypoxia times.

Changes in the value of the NIRS depends on 3 criteria: the tissue blood flow, the percentage of oxyhemoglobin and deoxyhemoglobin percentage.

ELIGIBILITY:
Inclusion criteria

* Children under 5 years
* Allowed in pediatric intensive care unit
* Having received heart surgery for management of congenital heart disease

Exclusion criteria

* Patients aged over 5 years
* Violations preexisting brain to the intervention (brain malformation)
* Patients with congenital heart disease and admitted to intensive care for reasons other than the surgical treatment of heart disease

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged under 5 years who underwent cardiac surgery (palliative or curative) and postoperative hospital period in pediatric resuscitation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
oxygen saturation in brain and kidney tissue | 1 hour after cardiac surgery

IPD SHARING:
Plan to Share IPD: No